CLINICAL TRIAL: NCT06668376
Title: A Study to Evaluate the Incrediwear Products Immediately After ACL or ACL+MCL Arthroscopic Surgery
Brief Title: A Study to Evaluate the Incrediwear Products Immediately After ACL Repair
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Bone and Joint (Other)
Collaborators: INCREDIWEAR HOLDINGS, INC. (Industry); Medical City Denton (Unknown)
Responsible Party: Principal Investigator, Christopher Flowers, MD, Orthopaedic Surgeon, Texas Bone and Joint
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRBNet 2205451-2
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Anterior Cruciate Ligament Tear; Medial Collateral Ligament
Keywords: Anterior Cruciate Ligament Tear; Medial Collateral Ligament Tear; Anterior Cruciate Ligament Repair; Medial Collateral Ligament Repair; Arthroscopic surgery
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: A Randomized Prospective Study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Placebo Product (Placebo Comparator): Once the informed consent has occurred, the patient will be invited to enroll in the study. The patient will be shown the Incrediwear products and given instructions. Participants will randomly be assigned treatment type in addition to the standard of care procedure they will be instructed to follow (active vs. placebo vs standard of care alone) based on surgery type. An equal number of patients from each primary condition type (ACL or ACL+MCL) will be assigned to each treatment type. The study will be double blinded as to the active vs placebo groups.
  Interventions: Device: Placebo
- Incrediwear Product (Active Comparator): Once the informed consent has occurred, the patient will be invited to enroll in the study. The patient will be shown the Incrediwear products and given instructions. Participants will randomly be assigned treatment type in addition to the standard of care procedure they will be instructed to follow (active vs. placebo vs standard of care alone) based on surgery type. An equal number of patients from each primary condition type (ACL or ACL+MCL) will be assigned to each treatment type. The study will be double blinded as to the active vs placebo groups.
  Interventions: Device: Leg Sleeve

INTERVENTIONS:
Device: Leg Sleeve — Once the informed consent has occurred, the patient will be invited to enroll in the study. The patient will be shown the Incrediwear product (Leg Sleeve) and given instructions. Participants will randomly be assigned treatment type in addition to the standard of care procedure they will be instructed to follow (active vs. placebo vs standard of care alone) based on surgery type. An equal number of patients from each primary condition type (ACL or ACL+MCL) will be assigned to each treatment type. The study will be double blinded as to the active vs placebo groups.
  Arms: Incrediwear Product
Device: Placebo — Once the informed consent has occurred, the patient will be invited to enroll in the study. The patient will be shown the Incrediwear product (Leg Sleeve) and given instructions. Participants will randomly be assigned treatment type in addition to the standard of care procedure they will be instructed to follow (active vs. placebo vs standard of care alone) based on surgery type. An equal number of patients from each primary condition type (ACL or ACL+MCL) will be assigned to each treatment type. The study will be double blinded as to the active vs placebo groups.
  Arms: Placebo Product

SUMMARY:
To assess the benefits of using the Incrediwear knee products after ACL or ACL+MCL arthroscopic surgery, on the postoperative pain, range of motion and effusion. The study team will compare patients with Incrediwear products, or placebo Incrediwear products, or no products during the first 6-month postoperative period. The group that does not wear the Incrediwear or placebo products is considered the standard of care control group and will proceed with the normal standard of care compression hose.

DETAILED DESCRIPTION:
After knee surgery, the participant will be randomly assigned to one of the three groups. The participant will have a 1-in-3 chance of being assigned to each group. The products will be placed on the participant by the hospital staff according to the random assignment sent with the surgical packet.

Study Screening/pre-operative appointment

* The surgeon confirms the participant meets the inclusion criteria and are scheduled for surgery in the next few weeks, and how the participant may be eligible to participate in the study.
* The surgeon will discuss the study and possible risks/benefits of being in the research.

  • Day of surgery
* The study packet will be sent to the hospital by the clinical staff. The packet will include a study number assignment, the products assigned the study number, and the patient study journal. The participant, surgeon, and hospital staff will not know which group the participant are in, with the exception of the standard of care control group, as this group will wear the hospital-issued compression hose.

  • Postoperative Recovery
* Subjective: Patient rates surgical site pain, on a 0-10 VAS pain scale. Patients will record pain medication type and quantity taken in a daily pain diary.
* Objective: Surgical extremity range of motion, and surgical extremity knee effusion, measured by either the Physical Therapist or the surgeon at the postop appointment.
* Measurements will be taken at; Preop appointment, Postop Day 0, Day 3, Day 7, Day 14, Day 21, Day 30 (1 month), Day 45, Day 60 (2 month), Day 100 (3 month), and Day 180 (6 month).

ELIGIBILITY:
Inclusion Criteria:

* Consented to protocol
* Compliant protocol
* BMI less than 35
* Undergoing ACL or ACL+MCL within 30 days

Exclusion Criteria:

* Pregnancy
* Rheumatoid Arthritis
* Poorly controlled diabetes (HgA1c > 7.5)
* Previous blood clots
* BMI greater than 35
* Varicosities on operative leg
* Pain management patient
* Prior knee surgery to the operative / study knee
* Worker's Comp patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2026-10-29 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | Preop appointment, Postop Day 0, Day 3, Day 7, Day 14, Day 21, Day 30 (1 month), Day 45, Day 60 (2 month), Day 100 (3 month), and Day 180 (6 month)
  The pain VAS is a unidimensional measure of pain intensity, used to record patients' pain progression, or compare pain severity between patients with similar conditions. The minimum number is zero meaning no pain and maximum number is 10 meaning the most pain the patient has every felt in their entire life. Lower scores are ideal while higher scores are indicative of the patient in a lot of pain.
Range of Motion Measured by a Goniometer | Preop appointment, Postop Day 0, Day 3, Day 7, Day 14, Day 21, Day 30 (1 month), Day 45, Day 60 (2 month), Day 100 (3 month), and Day 180 (6 month)
  Knee flexion and extension to assess mobility and functionality of the knee joint. The knee joint's range of motion (ROM) is an important clinical parameter used in knee assessment. Knee flexion should be about 150 degrees and knee extension should be about zero degrees (American Medical Association). Lower degrees of flexion are not ideal while higher degrees of extension are not optimal.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Flowers, MD, MS, Principal Investigator — Texas Bone and Joint
Locations (1):
- Medical City Denton, Denton, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Pre-approval to share data and data results must be obtained by the corporation.

REFERENCES:
- See also: Leg Sleeve — https://incrediwear.com/